CLINICAL TRIAL: NCT04258228
Title: Trans-coronary Pacing to Assess Myocardial Viability
Brief Title: Transcoronary Pacing and Myocardial Viability
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CD19/124706
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Cardiac Pacing, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Narrowing of the coronary arteries can cause chest pain and weaken the heart. In patients who have had heart attacks, blocked or severely narrowed arteries should be investigated (with coronary artery x-rays, or angiography) with efforts undertaken to improve the blood flow (angioplasty and stenting or heart bypass surgery). Sometimes these arteries are in fact supplying heart tissue which is already dead. Procedures to open up these vessels will therefore not influence how the patient feels or their future prognosis. On occasion, in order to determine whether heart tissue is alive (viable) and likely to benefit from of such efforts, a further investigation is required before another attempt is undertaken to open up these diseased arteries. This will require imaging of the heart to assess the state of the tissue (for example with magnetic resonance imaging, or cardiac MRI which is the gold standard). This means that patients may require two invasive procedures. One way around this would be to assess the electrical properties of the heart muscle in question during a single procedure. The principle is simply that dead muscle will have no electrical activity. Assessing the electrical properties of the heart through the coronary arteries using the same equipment used to treat the diseased artery during initial coronary angiography may provide viability information instantly, thus allowing treatment to proceed at the same procedure. In order to investigate whether this approach has promise, we will be performing a cardiac MRI around the time that patients have their coronary angioplasty. The electrical data will be compared to the cardiac MRI results to determine if this technique can be used in clinical practice. This innovative work has potential clinical and financial benefits.

Furthermore, patients can be diagnosed and treated during one procedure

ELIGIBILITY:
Inclusion Criteria:

- 1. Out Patients over 18 years who have been listed for electively for percutaneous coronary intervention.

2. In Patients who have been admitted with an acute coronary syndrome undergoing angiography query proceed

Exclusion Criteria:

* 1. Patients deemed to be in the terminal stage of illness; and patients who are unable to give informed consent.

  2. Atrial fibrillation with uncontrolled ventricular response at the time of procedure 3. The presence of a total occlusion of a coronary artery 4. Contra indications to coronary intervention 5. Patients with contraindications for cardiac MRI (See appendix) (15) 6. Patients with prior CABG 7. Patients who are claustrophobic 8. ST elevation myocardial infarction 9. Patients who have pace maker in situ 10. Patients on class I and III antiarrhythmics 11. Patients with haemodynamic instability

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified from elective waiting lists for percutaneous coronary interventions.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Transcoronary mapping | 60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom